CLINICAL TRIAL: NCT05672576
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy, Safety, and Tolerability of Cenerimod in Adult Subjects With Moderate-to-severe Systemic Lupus Erythematosus (SLE) on Top of Background Therapy
Brief Title: A Research Study to Evaluate the Efficacy and Safety of Cenerimod in Subjects Suffering From Systemic Lupus Erythematosus
Acronym: OPUS-2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Viatris Innovation GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ID-064A302; 2022-002815-47 (EudraCT Number); 2024-515871-37-00 (EU CTIS Number)
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-08

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Musculoskeletal and connective tissue disorders; Immune System Diseases; Autoimmune Diseases
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Connective Tissue Diseases; Immune System Diseases; Autoimmune Diseases | interventions — cenerimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cenerimod 4 mg (Experimental): Participants will receive cenerimod once daily in addition to background SLE therapy.
  Interventions: Drug: Cenerimod
- Placebo (Placebo Comparator): Participants will receive matching placebo once daily in addition to background SLE therapy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cenerimod — Cenerimod will be supplied as film-coated tablets at the dose of 4 mg.
  Other Names: ACT-334441
  Arms: Cenerimod 4 mg
Drug: Placebo — Matching placebo will be supplied as identical film-coated tablets formulated with the same excipients but without the active ingredient, cenerimod.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to see how well cenerimod reduces symptoms of Systemic Lupus Erythematous in adult patients with moderate to severe symptoms. The main questions it aims to answer are:

* How well cenerimod works on top of the treatment already being administered.
* How safe cenerimod is for adult patients with Systemic Lupus Erythematosus.

Researchers will compare one dose of cenerimod and a placebo to see how well cenerimod works when it is added to the treatment already being administered.

In this research study approximately 210 participants will receive cenerimod and approximately 210 participants will receive placebo for 12 months.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria at screening:

* Signed Informed Consent Form (ICF) prior to any study-mandated procedure.
* Diagnosis of Systemic Lupus Erythematosus (SLE) made at least 6 months prior to Screening, according to 2019 European League Against Rheumatism / American College of Rheumatology Criteria.
* A modified Systemic Lupus Erythematosus Disease Activity Index-2000 (mSLEDAI-2K) score ≥ 6 and clinical mSLEDAI-2K score ≥ 4 with at least 2 points for musculoskeletal or mucocutaneous manifestations (i.e., myositis, arthritis, rash, alopecia, mucosal ulcers). The mSLEDAI-2K score does not include "leukopenia".
* British Isles Lupus Assessment Group-2004 (BILAG) Grade B in ≥ 2 organ systems or a BILAG Grade A in ≥ 1 organ system.
* Physician's Global Assessment (PGA) score ≥ 1.0 on a 0 to 3 visual analog scale.
* Currently treated with one or more of the following SLE background medications:

  * Anti-malarials (≤ 400 mg/day hydroxychloroquine, ≤ 500 mg/day chloroquine, ≤ 100 mg/day quinacrine).
  * Mycophenolate mofetil (≤ 2 g/day) / mycophenolic acid (≤1.44 g/day).
  * Azathioprine (≤ 2 mg/kg/day).
  * Methotrexate (≤ 25 mg/week).
  * Oral Corticosteroids (OCS):

    * if OCS is the only SLE background medication: ≥ 7.5 mg/day and ≤ 30 mg/day prednisone or equivalent.
    * if OCS is not the only SLE background medication: ≤ 30 mg/day prednisone or equivalent.
  * Belimumab (≤10 mg/kg every 4 weeks intravenously [i.v.], or 200 mg/week subcutaneously [s.c.]).

Treatment with antimalarials, mycophenolate mofetil, mycophenolic acid, azathioprine, methotrexate or belimumab must have been started at least 90 days prior to Screening. Treatment with OCS must have been started at least 30 days prior to Screening.

• For women of childbearing potential (WoCBP):

* Negative serum pregnancy test at Screening.
* Agreement to undertake monthly urine pregnancy tests from Randomization up to 6 months after study treatment discontinuation.
* Agreement to use a highly effective method of contraception from Screening (Visit 1) up to 6 months after study treatment discontinuation.

Inclusion criteria at randomization:

* A clinical mSLEDAI-2K score ≥ 4 with at least 2 points for musculoskeletal or mucocutaneous manifestations (i.e., myositis, arthritis, rash, alopecia, mucosal ulcers).
* BILAG Grade B in 2 or more organ systems or a BILAG Grade A in 1 or more organ system.
* PGA score ≥ 1.0 on a 0 to 3 visual analog scale.
* Presence of at least one of the following biomarkers of serological evidence of active SLE (in a Screening sample as measured by central laboratory):

  * Anti-dsDNA antibodies elevated above normal,
  * Antinuclear antibodies with a titer of at least 1:160,
  * Anti-Smith antibody elevated above normal.
* Currently treated with one or more of the following SLE background medications that must be stable for at least 30 days prior to Randomization (except OCS, which must be stable for at least 15 days prior to Randomization):

  * Antimalarials (≤ 400 mg/day hydroxychloroquine, ≤ 500 mg/day chloroquine, ≤ 100 mg/day quinacrine);
  * Mycophenolate mofetil (≤ 2 g/day) / mycophenolic acid (≤ 1.44g/day);
  * Azathioprine (≤ 2 mg/kg/day);
  * Methotrexate (≤ 25 mg/week);
  * OCS:

    * if OCS is the only SLE background medication: ≥ 7.5 mg/day and ≤ 30 mg/day prednisone or equivalent.
    * if OCS is not the only SLE background medication: ≤ 30 mg/day prednisone or equivalent.
  * Belimumab (≤ 10 mg/kg every 4 weeks i.v. or ≤ 200 mg/week s.c.).
* WoCBP must have a negative urine pregnancy test at Randomization.

Main Exclusion Criteria:

* Pregnant, planning to be become pregnant up to Final Study Visit, or lactating women.
* Severe active central nervous system lupus or active severe or unstable neuropsychiatric SLE including but not limited to: aseptic meningitis; cerebral vasculitis; myelopathy; demyelination syndromes (ascending, transverse, acute inflammatory demyelinating polyradiculopathy); acute confusional state; impaired level of consciousness; psychosis; acute stroke or stroke syndrome; cranial neuropathy; status epilepticus; cerebellar ataxia; or mononeuritis multiplex:

  * That would make the subject unable to fully understand the ICF; OR
  * Where, in the opinion of the investigator/delegate, protocol-specified standard of care is insufficient and the use of a more aggressive therapeutic approach, such as adding i.v. cyclophosphamide and/or high dose i.v. pulse corticosteroid (CS) therapy or other treatments not permitted in the protocol is indicated.
* A diagnosis of mixed connective tissue disease or any history of overlap syndromes of SLE with psoriasis, rheumatoid arthritis, erosive arthritis, scleroderma, autoimmune hepatitis or uncontrolled autoimmune thyroid disease.
* History or presence of Mobitz type II or third-degree atrioventricular block, sick sinus syndrome, symptomatic bradycardia or syncope associated with cardiac disorders.
* Subjects who experienced myocardial infarction, unstable angina pectoris, stroke, transient ischemic attack, vascular thrombosis, decompensated heart failure requiring hospitalization, or heart failure defined by the New York Heart Association Class III/IV within 6 months prior to Screening.
* Resting heart rate < 50 bpm as measured by the 12-lead ECG at Screening or at Randomization.
* An elevated QT interval corrected according to Fridericia's formula (QTcF) interval of > 470 ms (females) / > 450 ms (males) at Screening or at Randomization.
* History or presence of severe respiratory disease or pulmonary fibrosis, based on medical history, lung function, and chest X-ray (or CT scan as per local guidelines), performed at Screening or within 6 months prior to Screening.
* History of clinically relevant bronchial asthma or chronic obstructive pulmonary disease that has required treatment with oral or parenteral CS for more than a total of 2 weeks within the last 6 months prior to Screening.
* History or presence of malignancy (except for surgically excised and non-recurrent cutaneous basal cell carcinoma, squamous cell carcinoma, or cervical carcinoma), lymphoproliferative disease, or history of total lymphoid irradiation within 10 years prior to Screening.
* Presence of any of the following abnormalities detected during the ophthalmological evaluation and/or by optical coherence tomography (OCT) during screening:

  * Macular edema of any cause: diabetic, cystoid, tractional.
  * Foveal degeneration, macular hole, macular pseudohole, hereditary or degenerative maculopathies.
  * Active uveitis, papilledema.
  * Retinal neovascularization of any cause and in any location.
* History of chronic liver or biliary disease (other than Gilbert's Syndrome) or subjects with alanine aminotransferase or aspartate aminotransferase > 3 × Upper Limit of Normal (ULN) or total bilirubin > 1.5 × ULN (unless in the context of known Gilbert's Syndrome).
* Significant hematology abnormality at screening assessment:

  * lymphocyte count < 500 /μL (0.5 × 10^9/L);
  * hemoglobin < 7 g/dL;
  * white blood cell count < 2000/μL (2.0 × 10^9/L); or
  * platelets < 25000/μL (25 × 10^9/L).
* Estimated glomerular filtration rate < 15 mL/min/1.73 m^2.
* Treatment with the following medications within 15 days or 5 half-lives of the medication (whichever is longer) prior to Randomization:

  * β-blockers, diltiazem, verapamil, digoxin, digitoxin, or any other antiarrhythmic or heart-rate -lowering systemic therapy.
  * QT-prolonging drugs with known risk of torsade de pointes irrespective of indication.
* Treatment with the following medications within 30 days or 5 half-lives of the medication (whichever is longer) prior to Randomization:

  * Cyclophosphamide, cyclosporine, voclosporin, tacrolimus, sirolimus, etc.
  * Pulse methylprednisolone.
  * Vaccination with live vaccines (including live vaccines for COVID-19).
* Intra-articular, intramuscular or i.v. CS within 6 weeks prior to Randomization.
* Treatment with the following medications within 90 days or 5 half-lives of the medication (whichever is longer) prior to Randomization:

  * Leflunomide.
  * i.v. immunoglobulins.
* Treatment with any investigational agent within 90 days or 5 half-lives of the drug (whichever is longer) prior to Randomization.
* Treatment with B cell-depleting biological agents (e.g., rituximab or ocrelizumab) or biological immunosuppressive agents (e.g., anti-tumor necrosis factor [TNF], anti-interleukin [IL]-1, anti-IL6 therapies), within 12 months prior to Randomization.
* Treatment with anifrolumab within 6 months prior to Randomization.
* Treatment with any of the following medications any time prior to Screening:

  * Alemtuzumab,
  * Sphingosine-1-phosphate receptor modulators (e.g., fingolimod),
  * Subjects previously randomized to cenerimod or placebo in any trial involving cenerimod.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Response on Systemic Lupus Erythematosus Responder Index 4 (SRI-4) at Month 12 compared to baseline | At Month 12 compared to Day 1 (pre-dose baseline)
  Response on SRI-4 is defined as:
  * Reduction from baseline of at least 4 points in the modified Systemic Lupus Erythematosus Disease Activity Index-2000 score (mSLEDAI-2K [SLEDAI-2K modified to exclude leukopenia, thus mSLEDAI-2K]), and
  * No new British Isles Lupus Assessment Group-2004 (BILAG) A organ domain score and not more than one new BILAG B organ domain score compared to baseline, and
  * No worsening from baseline in subjects' lupus disease activity, where worsening is defined as an increase ≥ 0.30 points on a 3-point Physician's Global Assessment visual analog scale (PGA VAS), and
  * No violation of specified medication rules detailed in the core protocol.

SECONDARY OUTCOMES:
Response on BILAG-based Composite Lupus Assessment (BICLA) at Month 12 compared to baseline | At Month 12 compared to Day 1 (pre-dose baseline)
  Response on BICLA is defined as:
  * Improvement from baseline in disease activity as measured by BILAG. Improvement is defined as a reduction of all baseline BILAG A to B/C/D and baseline BILAG B to C/D and no BILAG worsening in other organ systems, where worsening is defined as ≥ 1 new BILAG A or ≥ 2 new BILAG B, and
  * No worsening from baseline in mSLEDAI-2K, where worsening is defined as an increase from baseline of > 0 points in mSLEDAI-2K, and
  * No worsening from baseline in the patient's lupus disease activity, where worsening is defined as an increase of ≥ 0.30 points on a 3-point PGA VAS, and
  * No discontinuation of investigational product, and
  * No violation of specified medication rules detailed in the core protocol.
Time to first confirmation of a 4-month sustained modified Systemic Lupus Erythematosus Disease Activity Index-2000 (mSLEDAI-2K) response | Day 1 (pre-dose baseline) to Month 12
  A response is defined as a reduction of at least 4 points from baseline.
Time to first confirmation of a 4-month sustained response in mucocutaneous manifestations (i.e., rash, alopecia, mucosal ulcers) | Day 1 (pre-dose baseline) to Month 12
  Response is defined as:
  * No increase in the overall mSLEDAI-2K score excluding mucocutaneous manifestations, and
  * Remission (score of zero) from baseline in the mSLEDAI-2K score of mucocutaneous manifestations.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Viatris Innovation GmbH
Locations (147):
- United States (18):
  - Tucson Clinical Research Institute, LLC, Tucson, Arizona
  - UCSD Perlman Medical Offices, La Jolla, California
  - Amicis Research Center, Northridge, California
  - BioSolutions Clinical Research Center, Poway, California
  - Hope Clinical Trials, Inc., Coral Gables, Florida
  - Vital Pharma Research, Hialeah, Florida
  - Tectum Medical Research, Hollywood, Florida
  - Alloy Clinical Research, LLC, Kissimmee, Florida
  - Allied Biomedical Research Institute, Miami, Florida
  - D&H National Research Centers INC, Miami, Florida
  - Professional research Center INC, Miami, Florida
  - San Marcus Research Clinic, Inc., Miami Lakes, Florida
  - Tandem Clinical Research, Marrero, Louisiana
  - RB Wellness Clinic, Las Vegas, Nevada
  - Columbia University Medical Center, New York, New York
  - Precision Comprehensive Clinical Research Solutions, Colleyville, Texas
  - Texas Arthritis Center, El Paso, Texas
  - Northwest Houston Arthritis Center, Houston, Texas
- Chile (7):
  - Biomedica Research Group, Providencia
  - Sociedad Médica del Aparato Locomotor S. A., Providencia
  - Estudios G y C Ltda, Santiago
  - Enroll SpA, Santiago
  - Centro de Especialidades Medicas Vanguardia, Temuco
  - Clinical Research Chile SpA, Valdivia
  - Hospital San José de Victoria, Victoria
- Czechia (2):
  - iMedica s.r.o., Brno
  - Institute of Rheumatology Prague, Prague
- Georgia (15):
  - LTD "New Plasma Clinic", Batumi
  - Institute of Clinical Cardiology, Ltd, Tbilisi
  - LTD "Tbilisi Central Hospital", Tbilisi
  - National Institute of Endocrinology Ltd., Tbilisi
  - Tbilisi Heart and Vascular Clinic Ltd., Tbilisi
  - Aversi Clinic LTD, Tbilisi
  - Medi Club Georgia Ltd., Tbilisi
  - Tbilisi Institute of Medicine, Tbilisi
  - JSC Jerarsi Clinic, Tbilisi
  - Ltd. Mtskheta Street Clinic, Tbilisi
  - The First Medical Center Ltd., Tbilisi
  - Caucasus Medical Centre, Tbilisi
  - LLC "Innova", Tbilisi
  - LLC Raymann, Tbilisi
  - LTD "Tbilisi Heart Center", Tbilisi
- Germany (4):
  - Fraunhofer-Institut für Translationale Medizin und Pharmakologie ITMP, Frankfurt am Main
  - Universitätsklinikum Leipzig, Leipzig
  - Johannes Wesling Klinikum Minden, Minden
  - Universitätsklinikum Münster (UKM), Münster
- India (9):
  - Shalby Hospitals, Ahmedabad
  - Chennai Meenakshi Multispeciality Hospital Pvt. Ltd., Chennai
  - IPGME&R and SSKM Hospital, Kolkata
  - Jasleen Hospital, Nagpur
  - Chopda Medicare & Research Centre, Nashik
  - AIIMS New Delhi, New Delhi
  - Center for Rheumatic Diseases, Pune
  - Yashoda Hospital, Secunderabad
  - Nirmal Hospital Private Limited, Surat
- Malaysia (6):
  - Hospital Selayang, Batu Caves
  - Universiti Kebangsaan Malaysia - Medical Centre, Cheras
  - Hospital Tuanku Fauziah, Kangar, Kangar
  - University of Malaya Medical Centre, Kuala Lumpur
  - Sarawak General Hospital, Kuching
  - Hospital Sibu, Sarawak, Sibu
- Mexico (13):
  - Consultorio Particular Dr. Miguel Cortés Hernández, Cuernavaca
  - Centro Integral en Reumatologia SA de CV (CIRSA), Guadalajara
  - Morales Vargas Centro de Investigación S.C., León
  - Boca Clinical Trials Mexico, S.C., Mexico City
  - Centro de Investigación Clínica GRAMEL, S.C., Mexico City
  - Clinstile, S.A. de C.V., Mexico City
  - Centro Multidisciplinario para el Desarrollo Especializado de la Investigacion Clinica en Yucatan S.C.P. (CEMDEICY S.C.P.), Mérida
  - Accelerium, S. de R.L. de C.V., Monterrey
  - UBAM Unidad Biomédica Avanzada Monterrey, Monterrey
  - Oaxaca contra el Cáncer A.C, Oaxaca City
  - Centro de Estudios Clínicos de Querétaro S.C., Querétaro
  - Clinical Research Institute S.C., Tlalnepantla
  - PCR Toluca - Phylasis Clinical Research, Toluca
- Peru (13):
  - Unidad de Investigación en Medicina Interna y Enfermedades Críticas / Hogar Clínica San Juan de Dios, Cayma
  - Centro de Investigacion Clinica Inmunoreumatologia / ACQ Medic SAC, Jesús María
  - Centro de Investigación del Hospital Militar Central, Jesús María
  - Alberto Sabogal Sologuren National Hospital, Lima
  - Hospital Maria Auxiliadora, Lima
  - Unidad de Investigación de la Clinica International, San Borja
  - Instituto Peruano del Hueso y la Articulación S.A.C. (IPHAR), San Isidro
  - Clínica Anglo Americana, San Isidro
  - Servicios Reumatológicos SOMA E.I.R.L. / Clinica El Golf, San Isidro
  - Unidad de Investigación en Reumatología e Inmunología CSJB, San Juan de Lurigancho
  - Hospital Nacional Cayetano Heredia, San Martín de Porres
  - Investigaciones Clinicas / Instituto de Ginecología y Reproducción, El Derby, Santiago de Surco
  - Centro de Investigación Clínica Trujillo EIRL / Clínica Peruano Americana S.A, Trujillo
- Philippines (6):
  - Iloilo Doctors Hospital, Iloilo City
  - Makati Medical Center, Makati
  - Ospital ng Makati, Makati City
  - St Lukes Medical Center, Manila
  - The Medical City Clark, Pampanga
  - St Luke's Medical Center Quezon City / University of Santo Tomas Hospital, Sampaloc
- Poland (6):
  - Szpital Uniwersytecki nr 2 im. dr. Jana Biziela w Bydgoszczy, Bydgoszcz
  - Santa Sp. z o.o., Lodz
  - Medyczne Centrum Hetmańska, Poznan
  - Twoja Przychodnia Poznańskie Centrum Medyczne, Poznan
  - Pomorski Uniwersytet Medyczny w Szczecinie, Szczecin
  - MICS Centrum Medyczne Warszawa, Warsaw
- Portugal (7):
  - Hospital Prof. Doutor Fernando Fonseca, Amadora
  - Centro Hospitalar Universitário do Algarve - Hospital de Faro, Faro
  - ULS Guarda, Guarda
  - Hospital Senhora Oliveira-Guimaraes, Guimarães
  - Instituto Portugues De Reumatologia, Lisbon
  - Unidade Local De Saude Lisboa Ocidental E.P.E., Lisbon
  - Centro Hospitalar de Vila Nova de Gaia/Espinho, E.P.E., Vila Nova de Gaia
- Puerto Rico (2):
  - Centro Reumatologico de Caguas, Caguas
  - GCM Medical Group, PSC, San Juan
- Serbia (8):
  - Institute of Rheumatology, Belgrade (study site 1), Belgrade
  - Institute of Rheumatology, Belgrade (study site 2), Belgrade
  - Institute of Rheumatology, Belgrade (study site 3), Belgrade
  - University Clinical Center of Serbia, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical Center Kragujevac, Kragujevac
  - Special Hospital for Rheumatic Diseases, Novi Sad, Novi Sad
  - General Hospital "Djordje Joanovic", Zrenjanin
- South Africa (5):
  - Arthritis Clinical Research Trials, Cape Town
  - Panorama Medical Centre, Cape Town
  - Charlotte Maxeke Johannesburg Academic Hospital, Parktown
  - University of Pretoria, Pretoria
  - Winelands Medical Research, Somerset West
- Spain (12):
  - Accellacare, Alcobendas
  - Parc Tauli Sabadell University Hospital, Barcelona
  - Hospital Universitari Vall d'Hebron, Colmenar Viejo
  - Hospital Universitario Ramon y Cajal, Colmenar Viejo
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Clinica Gaias Santiago, Santiago de Compostela
  - Hospital QuironSalud Sagrado Corazon, Seville
  - Hospital Universitario Nuestra Señora de Valme, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitario Doctor Peset, Valencia
  - Hospital Universitario Río Hortega de Valladolid, Valladolid
- Ukraine (12):
  - Communal Non-profit Enterprise "Chernihiv Regional Hospital" of the Chernihiv Regional Council, Rheumatology Department, Chernihiv
  - St. Luke's Treatment and Diagnostic Center, Ivano-Frankivsk
  - Medical Center "Harmoniia krasy", LLC, Kyiv
  - Medical Center of the Limited Liability Company "Edelweiss Medics", Treatment and Prevention Department, Kyiv
  - Med Center "Ok!Clinic+" of Ltd Liability Com "Inter Ins of Clin Rsrch", Inpatient dprt, Unit of Ther, Rheuma and Cardio, Kyiv
  - "Medbud-Clinic" LLC, Treatment and Prevention Department of the Medical Center, Kyiv
  - Medical Center "Universal Clinic "Oberih"" of Limited Liability Company "Capital", Kyiv
  - Limited Liability Company "Medical Centre 'Consilium Medical'", Clinical and Consultation Department, Kyiv
  - Medical Center "Center of Family Medicine Plus" LLC, Treatment and Prevention Department, Kyiv
  - Ternopil Regional Clinical Hospital, Ternopil
  - "Medical Center Health Clinic" LLC, Medical Clinical Investigational Center, Department of Cardiology and Rheumatology, Vinnytsia
  - Communal Non-Com Entr Vinnytsia City Clin Hpt 1, Clin Therapy Dprt 2, Vinnytsia Nat Pirogov Memo Med Uni, Dprt of Internal Med 3, Vinnytsia
- United Kingdom (2):
  - University Hospitals of Leicester Nhs Trust, Leicester
  - Guy's and St. Thomas' NHS Foundation Trust - Guy's Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Askanase AD, D'Cruz D, Kalunian K, Merrill JT, Navarra SV, Cahuzac C, Cornelisse P, Murphy MJ, Strasser DS, Trokan L, Berkani O. Cenerimod, a sphingosine-1-phosphate receptor modulator, versus placebo in patients with moderate-to-severe systemic lupus erythematosus (CARE): an international, double-blind, randomised, placebo-controlled, phase 2 trial. Lancet Rheumatol. 2025 Jan;7(1):e21-e32. doi: 10.1016/S2665-9913(24)00246-7. Epub 2024 Nov 22. PMID 39586304